CLINICAL TRIAL: NCT07346859
Title: Open-label, Multicentre, Tolerability, Safety and Pharmacokinetics Study of the Medicinal Product BP-SCIG 20% (Human Normal Immunoglobulin for Subcutaneous Administration) Manufactured by BIOPHARMA PLASMA LLC, Followed by an Efficacy Assessment of Long-term Use in Patients With Primary Immunodeficiency (PID)
Brief Title: Study of BP-SCIG 20% in Patients With Primary Immunodeficiency (PID)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biopharma Plasma LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SCIg-BP
Record Dates: First submitted 2025-12-26; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Primary Immunodeficiency Diseases
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: This study does not involve the distribution of patients into groups. Of patients in all age categories who meet inclusion criteria and passed the screening, and who do not meet any of the non-inclusion (exclusion) criteria, one group is formed, which will receive the investigational product.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group receiving BP-SCIG20% (Experimental): Patients receive BP-SCIG 20% (human normal immunoglobulin, 200 mg/mL, IgG ≥95%) administered subcutaneously. Dosage: 0.4-0.8 g/kg per month, divided into weekly infusions. Duration: Long-term treatment as per study protoco
  Interventions: Drug: BP-SCIG 20%

INTERVENTIONS:
Drug: BP-SCIG 20% — Human normal immunoglobulin 200 mg/mL (including immunoglobulin G (IgG) no less than 95 %) administered subcutaneously.
  Distribution of immunoglobulin G subclasses in the product:
  IgG1: 65.6 %, IgG2: 22.1 %, IgG3:10.8 %, IgG4:1.5 % The maximum content of immunoglobulin A is 100 µg/mL.

SUMMARY:
All patients will receive the investigational medicinal product BP-SCIG 20%, solution for subcutaneous administration, manufactured by BIOPHARMA PLASMA LLC. A loading dose of IMP may be required (at the Investigator's decision): at least 0.2-0.5 g/kg (1.0-2.5 mL/kg) of body weight. This dose is distributed across several days, with a maximum daily dose of 0.1 to 0.15 g/kg. After achieving a steady-state (minimal) level of IgG, maintenance doses are administered at repeated intervals (approximately once a week) to achieve a cumulative monthly dose of 0.4-0.8 g/kg.

DETAILED DESCRIPTION:
The clinical trial will consist of three periods, namely:

screening period: lasting up to 2 months, and involving three screening visits; treatment period (from Cycle 1 visit [the first 4 administrations of the IMP are to be performed in a hospital setting] during the 52 weeks to the last visit of Cycle 13).

follow-up period after completion of the last cycle of the treatment period, with a duration of 1 week.

ELIGIBILITY:
Inclusion Criteria:

* a signed informed written consent of the patient/patient's parents or legally authorised representative to take part in the study;
* children from 0 to 18 years of age, of both sexes; or adult patients: males and females older than 18 years;
* a diagnosis of primary immunodeficiency with impaired antibody production document-supported according to the ESID criteria, requiring replacement therapy with immunoglobulins;
* patients with a body weight of no less than 9.1 kg;
* patients who received replacement therapy with intravenous immunoglobulin (IVIG) products at intervals from 21 to 28 days at the dose of 0.4-0.8 g/kg, for at least 4 months prior to the start of the study and have total serum IgG levels ≥5 g/L*, which is confirmed by the results of no less than 2 measurements performed immediately before the scheduled IVIG administration after signing the ICF, or patients who received replacement therapy with subcutaneous immunoglobulin (SCIG) products at the dose of 0.4-0.8 g/kg per month, for at least 4 months prior to the start of the study, and have total serum IgG levels ≥5 g/L*, based on the results of no less than 2 measurements performed immediately before the scheduled SCIG administration after signing the ICF; or patients with a newly established diagnosis of PID who have not yet received replacement therapy with IgG products (treatment-naïve patients) and have a serum IgG level ≤ 4 g/L;
* absence of episodes of serious bacterial infections (bacteraemia or sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, visceral abscess) while taking the previous medicinal product and absence of episodes of hospitalisation for at least 3 months prior to inclusion in the study and during the screening period (prior to the first administration of the IMP BP-SCIG 20%);
* a negative pregnancy test (in female patients with childbearing potential); readiness to use reliable methods of contraception throughout the study period;
* patient's ability, in the Investigator's judgement, to comply with all the requirements of the study protocol.

Exclusion Criteria:

* at the request of the patient/patient's parents/patient's legally authorised representative at any time and for any reason;
* patient developing serious and/or unexpected AEs/ARs during the study, which require discontinuation of the product;
* blood transfusions or transfusions of blood components and products, with the exception of the IMP;
* the need to use medicinal products disallowed as part of this study;
* systematic lack of patient compliance with the treatment regimen prescribed by the Investigator;
* systematic lack of patient compliance with the procedures specified in this protocol;
* exclusion based on screening results, including emergence of episodes of serious bacterial infections while receiving a previous IV immunoglobulin product and episodes of hospitalisation during the screening period (before the first administration of the IMP BP-SCIG 20%).
* Receiving the IMP BP-SCIG 20% for less than 4 months;
* Presence of episodes of serious bacterial infections (bacteraemia or sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, visceral abscess) at the time of investigation of PK parameters.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Trough Plasma Concentration of Total IgG at Steady State | From baseline through 12 months of treatment
  Mean monthly trough plasma concentration of total IgG prior to the next BP-SCIG 20% infusion, measured after 4 months of treatment and assessed over 6 months, compared with previous therapy (BIOVEN).
Number of Serious Bacterial Infections per Subject per Year | From baseline through 12 months of treatment
  Occurrence of less than 1 serious bacterial infection per patient per year during 52 weeks of BP-SCIG 20% treatment. Serious bacterial infection includes sepsis, bacterial pneumonia, bacterial visceral infections, bacterial meningitis, osteomyelitis/septic arthritis.

SECONDARY OUTCOMES:
Fraction of patients reaching IgG ≥5 g/L | From baseline through 12 months of treatment
  Percentage of patients achieving serum IgG ≥5 g/L prior to scheduled infusion.
Incidence of non-serious infections | From baseline through 12 months of treatment
  Number of non-serious infectious disease episodes per patient per year
Duration of non-serious infections | From baseline through 12 months of treatment
  Total duration of non-serious infections per patient per year.
Antibiotic use | From baseline through 12 months of treatment
  Fraction of patients receiving antibiotics and mean number of days of antibiotic therapy per year.
Hospital admissions due to infection | From baseline through 12 months of treatment
  Number and duration of hospital admissions due to infection per patient per year.

CONTACTS AND LOCATIONS:
Locations (12):
- Ukraine (12):
  - Municipal Non-Profit Enterprise "Cherkasy Regional Children's Hospital" of the Cherkasy Regional Council, Cherkasy
  - Regional Municipal Non-Profit Enterprise "Chernivtsi Regional Teaching Hospital", Chernivtsi
  - Municipal Non-Profit Enterprise "Ivano-Frankivsk Regional Teaching Hospital" of the Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Municipal Non-Profit Enterprise "Ivano-Frankivsk Regional Children's Teaching Hospital" of the Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Municipal Non-Profit Enterprise "Kyiv City Children's Teaching Hospital No. 1", Kyiv
  - LLC "Allergy and Cough Clinic", Lutsk
  - Municipal Enterprise "Volyn Regional Territorial Medical Association for the Protection of Motherhood and Childhood" of the Volyn Regional Council, Lutsk
  - Municipal Non-Profit Enterprise of the Lviv Regional Council "Lviv Regional Teaching Diagnostic Centre", Lviv
  - Municipal Non-Profit Enterprise of the Lviv Regional Council "Clinical Centre of Children's Medicine", structural unit "West Ukrainian Specialised Centre", Lviv
  - Municipal Non-Profit Enterprise "Central Municipal Hospital" of Rivne City Council, Rivne
  - Municipal Non-Profit Enterprise "Vinnytsia Regional Teaching Hospital named after M.I. Pyrohov" of the Vinnytsia Regional Council, Vinnytsia
  - Municipal Non-Profit Enterprise "Vinnytsia Regional Children's Teaching Hospital" of the Vinnytsia Regional Council, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT07346859/Prot_000.pdf